CLINICAL TRIAL: NCT04677686
Title: Observation of the Implementation of a Bundle of Care in Colorectal Surgery to Reduce Surgical Site Infections Successfully
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Other Study IDs: 220-00051
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Reduction of Surgical Site Infections in Colorectal Surgery
Keywords: colorectal surgery; bundle of care; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-implementation phase (October 2018 - September 2019): During this time period, 137 patients underwent colorectal surgery. Only basic measures for preventing SSI were performed:
  1. Hair was removed in the operating field with a clipper instead of shaving hair.
  2. Blood glucose was monitored only during the operation.
  3. Antibiotic prophylaxis was applied 60 minutes before the operation.
  4. The application of an antibiotic prophylaxis was repeated if the operation lasted longer than 4 hours.
  5. Measures of warming were only applied during the operation and in the recovery room.
  6. Instruments and gloves were changed after finishing the anastomosis.
- Implementation phase (October 2019 - September 2020): During this phase, additional measures have been introduced:
  1. Implementation of wound protectors during colorectal surgery.
  2. Colorectal operations were only performed with the support of an experienced consultant surgeon.
- Post-implementation phase (October 2020 - September 2021): During this phase, additional measures are implemented.
  1. Close monitoring of blood glucose. During the stay in the recovery room and for 48 hours post-operative, blood glucose is monitored closely. Moreover, if blood glucose is higher than 9 mmol/l, the patient will be treated with insulin. This measure is applied to diabetic as well as to non-diabetic-patients.
  2. The measures of warming will be intensified. First of all, during the operation and during the stay in the recovery room patients will be placed on warming mattresses. Moreover, a warming towel will be placed on the operating field directly after the operation.
  3. The patients will be asked to take a shower the night before surgery. In case of an emergency operation, patients will be asked to wash the axilla, trunk, genitalia, groins and umbilicus
  Interventions: Behavioral: Bundle of Care

INTERVENTIONS:
Behavioral: Bundle of Care — Hair removal with Clipper Glucose Control Preoperative antibiotics Repeat antibiotics after 4 Hours Optimize Body temperature Instrument change for colorectal anastomosis Use of wound protectors Experienced surgeon Preoperative showering
  Groups: Post-implementation phase (October 2020 - September 2021)

SUMMARY:
This study aims to evaluate whether the colorectal bundle designed and implemented at Cantonal Hospital Lucerne, will lead to a significant reduction of SSIs. The impact of potential risk factors for SSIs will additionally be evaluated.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) remain a relevant problem in colorectal surgery. The aim of this study is to implement a bundle of care in order to reduce SSIs in colorectal surgery.

All patients undergoing colorectal surgery between October 2018 and September 2021 will be included in a prospective observational study. Since our colorectal bundle has been established gradually, patients will be grouped in a pre-implementation (2018-2019), implementation (2019-2020) and post implementation phase (2020-2021), in order to assess the effectiveness of the actions undertaken. Primary endpoint of this study will be surgical site infection (SSI) rate, while secondary endpoints encompass potential risk factors for SSIs. We assume that obesity, age, diabetes, alcoholism and smoking may lead to a higher risk for SSIs.

ELIGIBILITY:
Inclusion Criteria:

over 18 elective or emergency colorectal surgery written informed consent

Exclusion Criteria:

pregnant no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal surgery in the Cantonal Hospital of Lucerne October 2020-September 2021
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Site infection | 30 days
  rate of SSIs and classification of SSIs (superficial SSI, deep SSI or organ space SSI)

SECONDARY OUTCOMES:
Risk factors for SSI | at surgery
  Determination of the risk factors for SSI (Obesity, age, diabetes, alcoholism, immune-deficit illnesses (such as HIV and Hepatitis), smoking, immunosuppressive drugs, chemotherapy, radiotherapy, COPD, pAVK, renal insufficiency and poor Nutrition)

CONTACTS AND LOCATIONS:
Overall Officials: Jörn-Markus Gass, Principal Investigator — Cantonal Hospital of Lucerne, Spitalstrasse, 6000 Lucerne 16
Locations (1):
- Cantonal Hospital of Lucerne, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brunner S, Liesenberg J, Fourie L, Metzger J, Scheiwiller A, Zschokke I, Lehnick D, Gass JM. Implementation of a Bundle of Care in Colorectal Surgery to Reduce Surgical Site Infections Successfully at Cantonal Hospital Lucerne: Study Protocol for a Prospective Observational Study. Int J Surg Protoc. 2021 Sep 23;25(1):220-226. doi: 10.29337/ijsp.150. eCollection 2021. PMID 34616960